CLINICAL TRIAL: NCT02576821
Title: Hippocampal Sclerosis and Amnesia Not Due to Alzheimer's Disease
Acronym: ShaTau7
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: D14-P010
Record Dates: First submitted 2015-10-13; First posted 2015-10-15 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Patients With Cognitive Disturbances
Keywords: Amnesia, Alzheimer, hippocampal sclerosis, fronto-temporal lobar degeneration
MeSH Terms: conditions — Amnesia; Hippocampal Sclerosis | interventions — Restraint, Physical

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Patients with Hippocampal sclerosis non AD (Other): Patients with Hippocampal sclerosis non AD (n=40)
  Interventions: Other: Neurological examinations; Other: Neuropsychological examinations; Other: Clinical examinations; Radiation: MRI 3T; Radiation: MRI 7T
- Patients with Alhzeimer's Disase (Other): Patients with Alhzeimer's Disase (n=40)
  Interventions: Other: Neurological examinations; Other: Neuropsychological examinations; Other: Clinical examinations; Radiation: MRI 3T; Radiation: MRI 7T
- Patients with DLFT (Other): Patients with DLFT (n=20)
  Interventions: Other: Neurological examinations; Other: Neuropsychological examinations; Other: Clinical examinations; Radiation: MRI 3T; Radiation: MRI 7T
- Patients with CBD/PSP (Other): Patients with CBD/PSP (n=20)
  Interventions: Other: Neurological examinations; Other: Neuropsychological examinations; Other: Clinical examinations; Radiation: MRI 3T; Radiation: MRI 7T
- Normal controls (Other): Normal controls (n=20)
  Interventions: Other: Neurological examinations; Other: Neuropsychological examinations; Other: Clinical examinations; Radiation: MRI 3T; Radiation: MRI 7T

INTERVENTIONS:
Other: Neurological examinations
Other: Neuropsychological examinations
Other: Clinical examinations
Radiation: MRI 3T
Radiation: MRI 7T

SUMMARY:
Hippocampal Sclerosis (HS) leads to anterograde amnesia mimicking early Alzheimer's disease (AD) (so called HSA-nonAD). Recent studies showed that (a) the deficit of episodic memory as well as the level of hippocampal atrophy in bvFTD may be of similar severity to that observed in AD, even at initial presentation, leading to misdiagnosis in 22% of cases with post mortem diagnosis; (b) amnesia with HS due to microvascular lesion and microinfarcts can also cause impairment of episodic memory mimicking AD, without subcortical cognitive profile. Because these diseases involve distinct pathophysiological processes, they require different specific care and treatment. In consequence, it is very important to improve our knowledge about HS in order to identify its mechanism and improve the diagnosis.

DETAILED DESCRIPTION:
Hippocampal sclerosis (HS) refers to neuronal cell loss and astrocytosis in subiculum and cornu ammonis subfields of the hippocampal formation unrelated to Alzheimer's disease pathology. In contrast to HS that affects younger adults with epilepsy, older individuals with HS have significant ante-mortem cognitive dysfunction but no epilepsy. Neuropathological studies demonstrated three main types of HS associated with aging: (a) HS-Ageing to refer to the disease with HS pathology in ageing individuals, observed in more than 10% of subjects aged over 85 years; (b) HS observed in the behavioural variant of frontotemporal dementia (bvFTD), HS being more frequent in tau-negative pathology, especially in FTLD-TDP. bvFTD patients may manifest severe episodic memory impairment and hippocampal atrophy; (c) HS associated with cortical or subcortical cerebral microinfarcts, which are invisible on conventional MRI. Cerebral microinfarcts are observed in 33% of elderly over 85 years in post-mortem studies.

HS leads to anterograde amnesia mimicking early Alzheimer's disease (AD) (so called HSA-nonAD). Recent studies showed that (a) the deficit of episodic memory as well as the level of hippocampal atrophy in bvFTD may be of similar severity to that observed in AD, even at initial presentation, leading to misdiagnosis in 22% of cases with post mortem diagnosis; (b) amnesia with HS due to microvascular lesion and microinfarcts can also cause impairment of episodic memory mimicking AD, without subcortical cognitive profile. Because these diseases involve distinct pathophysiological processes, they require different specific care and treatment. In consequence, it is very important to improve our knowledge about HS in order to identify its mechanism and improve the diagnosis.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria

* Be older than18 years old.
* Consulting in one of the centers (patients only)
* Sufficient cognitive capacities for the realization of the clinical and neuropsychological evaluations, left to the judgement by the investigator.
* Women old enough to procreate under effective contraception
* Signed consent
* Absence of general or systemic disorders that may interfere with cognition.
* If available before inclusion, absence of brain lesions as determined by MRI that may account for even part of the clinical presentation.

Patients with Hippocampal sclerosis non AD (n=40)

Clinical criteria :

* CDR (Clinical Dementia Rating Scale) = 0.5 or 1
* Progressive amnestic syndrome of the hippocampal type, defined by a free recall score ≤ 17/48 and a total recall score ≤ 40/48 on the FCSRT.

Biological criteria : Absence of Profile suggestive of AD on the study of the biomarkers of the CSF (IATI ratio > 0.8)

Patients with Alheimer's Disase (n=40)

Clinical criteria :

* CDR (Clinical Dementia Rating Scale) = 0.5 or 1
* Typical amnesic AD : Progressive amnestic syndrome of the hippocampal type, defined by a free recall score ≤ 17/48 and a total recall score ≤ 40/48 on the FCSRT, associated or not with others cognitive impairment
* Posterior Cortical Atrophy : initial presentation of progressive visual or visuospatial impairment; absence of ophthalmologic impairment with evidence of complex visual and/or visuospatial disorder on examination; a relatively preserved episodic memory
* Logopenic progressive aphasia : word retrieval deficits in spontaneous speech and confrontation naming, impaired repetition of sentences, errors in spontaneous speech and naming (eg, phonological errors), and relative sparing of word and object knowledge and motor speech.

Biological criteria : CSF biomarkers suggestive of AD defined on CSF.

Patients with DLFT (n=20) :

Clinical criteria :

* Modifications of the personality and the social conducts in the foreground
* Compatible brain imaging with the diagnosis : profile of atrophy and/or hypometabolism in TEP-FDG (or hypoerfusion in Spect) compatible with the diagnosis of DFT and/or absence of atypie Biological criteria : No AD profile on CSF biomarkers

Patients with CBD/PSP (n=20) (Armstrong et al., 2013)

1. Corticobasal syndrome :

   * at least one of the following signs : limb rigidity or akinesia, limb dystonia, limb myoclonusplus at least one of the following sign : orobuccal or limb apraxia, e) cortical sensory deficit, alien limb phenomena (more than simple levitation)
   * Nonfluent/agrammatic variant of primary progressive aphasia: Effortful, agrammatic speech plus at least one of: a) impaired grammar/sentence comprehension with relatively preserved, single word comprehension, or b) groping, distorted speech production (apraxia of speech)
2. Progressive supranuclear palsy syndrome :

   * Three of the following items present: a) axial or symmetric limb rigidity or akinesia, b) postural instability or falls, c) urinary incontinence, d) behavioural changes, e) supranuclear vertical gaze palsy or decreased velocity of vertical saccades

Normal controls (n=20):

Absence of known psychiatric disorder Score on the Folstein Mini Mental Status (MMSE > or = 27) Normal neuropsychological assessment for the age and the educational level

Exclusion Criteria:

* Subject with a psychiatric evolutionary and/or badly checked pathology (left to the judgement of the investigator).
* Subject with a grave, severe or unstable pathology (left to the judgement of the investigator) the nature of which can interfere with the variables of evaluation.
* Epileptics subjects, badly tolerant MRI (1.5T, 3T or 7T), Subject presenting contraindications to the MRI (if necessary, a blood pregnancy test will be performed before 7T MRI) (Pacemaker or stimulating neurosensory or implantable defibrillator, cochlear implants, eye or cerebral ferromagnetic foreign bodies close to nervous structures, metallic prostheses, agitation of the patient : not cooperative or agitated patients, very young children, claustrophobics subjects, pregnant women, neurosurgical ventriculoperitoneal shunt valves, brace)
* Known or supposed histories (< or = 5 years) of severe alcoholism or misuse of drugs
* Vascular, inflammatory or expansive, visible lesion in the MRI which can interfere on the criteria of diagnosis.
* No health insurance
* Pregnant, breast-feeding woman or planning a pregnancy in two years of follow-up.
* For controls : anomaly detected on the MRI in the appreciation of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
7 tesla MRI. | up to Month 18
  Structural morphometric analysisze of hippocampal and Papez circuit sub-regions, and detection of microinfarcts/microbleeds by 7 tesla MRI.

SECONDARY OUTCOMES:
3T MRI | Baseline
  Morphometry of hippocampus by 3T MRI
3T MRI | Month 12
  Morphometry of hippocampus by 3T MRI
3T MRI | Month 24
  Morphometry of hippocampus by 3T MRI
3T MRI | Baseline
  White matter intensities assessed by 3T MRI
3T MRI | Month 12
  White matter intensities assessed by 3T MRI
3T MRI | Month 24
  White matter intensities assessed by 3T MRI
7T MRI | up to Month 18
  Volumetry of the cholinergic nucleus basalis by 7T MRI
CSF | Baseline
  CSF biomarkers
Neuropsychological assessment | Baseline
  Neuropsychological assessment
Neuropsychological assessment | Month 12
  Neuropsychological assessment
Neuropsychological assessment | Month 24
  Neuropsychological assessment
Clinical assessment | M0
  Clinical assessment
Clinical assessment | Month 12
  Clinical assessment
Clinical assessment | Month 24
  Clinical assessment
Genetic markers of bvFTD | Baseline
  Genetic markers of bvFTD
Blood markers | Baseline
  Blood markers
Plasmatic progranulin levels | Baseline
  Plasmatic progranulin levels
Regional glucose hypometabolism | Baseline
  Regional glucose hypometabolism assessed by FDG-PET (if performed during clinical care).

CONTACTS AND LOCATIONS:
Overall Officials: Marie SARAZIN, MD, PhD, Principal Investigator — Centre Hospitalier Sainte-Anne
Locations (1):
- Neurologie de la mémoire et du langage, Service de Neurologie, Centre Hospitalier Sainte-Anne, Paris, France